CLINICAL TRIAL: NCT02982590
Title: Apixaban Versus Warfarin in Patients With Left Ventricular Thrombus: A Prospective Randomized Outcome Blinded Study on the Size Reduction or Resolution of Left Ventricular Thrombus
Brief Title: Apixaban Versus Warfarin in Patients With Left Ventricular Thrombus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Institut Jantung Negara (Other)
Responsible Party: Principal Investigator, Dr W. Yus Haniff W. Isa, DR, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 304/PPSP/61313197
Record Dates: First submitted 2016-11-21; First posted 2016-12-05 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Left Ventricular Thrombosis
MeSH Terms: interventions — apixaban; Tablets; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- warfarin sodium (Active Comparator): warfarin daily, dosage according to INR monitor. Aim INR 2-3
  Interventions: Drug: Warfarin Sodium
- apixaban (Experimental): Apixaban 5 MG Oral Tablet [ELIQUIS] will be given for randomly selected patients for 3 months.
  Interventions: Drug: Apixaban 5 MG Oral Tablet [ELIQUIS]

INTERVENTIONS:
Drug: Apixaban 5 MG Oral Tablet [ELIQUIS] — Apixaban is licensed for treatment of deep vein thrombosis and pulmonary embolism. Hence, a good study drug for left ventricular thrombosis for possibility of a new indication.
  Other Names: ELIQUIS
  Arms: apixaban
Drug: Warfarin Sodium — as controlled arm since warfarin is the standard therapy for LV thrombus
  Other Names: Coumadin
  Arms: warfarin sodium

SUMMARY:
The purpose of this study is to compare the novel oral anticoagulant apixaban with the standard therapy of warfarin on the size reduction or resolution of left ventricular thrombus over 3 months.

DETAILED DESCRIPTION:
Current treatment for left ventricular thrombus is anti-coagulant or blood thinning agent known as warfarin. Recently at least three novel oral anticoagulant agents were used in the treatment of atrial fibrillation, pulmonary embolism and deep vein thrombosis (DVT).

Novel oral anticoagulant drugs will require no blood taking for INR monitoring, hence less visit and more convenience to patients. Latest studies also showed lesser rate of bleeding as compared to warfarin and hence relatively safer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80 years old
2. Presence of LV thrombus or spontaneous echo contrast (SEC) grade 3 or 4 (Patel VG 1996), with regional wall motion abnormalities
3. HASBLED score less than 3
4. No episodes of major bleeding in the past 6 months a) Major bleeding defined as i. episodes of bleeding with significant drop in haemoglobin(Hb)level of at least 2gm/dL - Includes upper and lower gastrointestinal bleed ii. The need for blood transfusion (pack cell) of at least 2 unit iii. Recent surgery with bleeding complications and lost of Hb as in (i) or (ii) iv. Any intracranial bleeds with neurological deficits

Exclusion Criteria:

1. Patient with unstable arrhythmias and/or recurrent cardiogenic shock
2. Patient with large ischemic stroke on recruitment-defined as involving >1/3 of cerebral hemisphere or deemed to have high chance of haemorrhagic transformation
3. Patient with permanent pacemaker
4. Patient who is post valve replacement therapy
5. Patient who is pregnant.
6. Patient with advanced kidney disease at stage V and not on dialysis (CrCl <15 mL/min)
7. Patient with advanced liver disease with coagulopathy
8. Patient with organized and old left ventricular thrombus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr W. Yus Haniff W. Isa, M.MED, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelanatan, Malaysia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Warfarin Sodium | Apixaban
Started | 13 | 14
Completed | 9 | 13
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 4 | 0

BASELINE CHARACTERISTICS:
Population: Gender, Age, Co-morbidities, HAS-BLED score
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin Sodium | Apixaban | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.00 (11.42) | 55.36 (11.04) | 55.19 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Comorbidities [Count of Participants; unit: Participants]
  Diabetes mellitus | 9 | 7 | 16
  Hypertension | 9 | 8 | 17
  Ischemic heart disease | 8 | 9 | 17
  Atrial fibrillation | 0 | 1 | 1
  Chronic kidney disease | 7 | 5 | 12
  Hyperlipidemia | 9 | 8 | 17
HAS-BLED score [Mean (Standard Deviation); unit: total score] — Hypertension, Abnormal renal or liver function, Stroke, Bleeding, Labile INR, Elderly, Drugs or alcohol (HAS-BLED) score estimates the 1-year risk of major bleeding for patients on anticoagulation to assess risk-benefit in atrial fibrillation care. Minimum score = 0, maximum score = 9.
  Score of 0 to 1: Low risk for major bleeding. Score of 2: Moderate risk for major bleeding. Score ≥ 3: High risk for major bleeding.
  In our study, we exclude patients with HAS-BLED score > 3. Thus, only patients with HAS-BLED score from 0 to 3 were recruited.
  total score | 1.46 (0.66) | 1.0 (0.68) | 1.22 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Left Ventricular Thrombus (LVT) Size
Description: Percentage of change in left ventricular thrombus (LVT) size after 12 weeks of Warfarin or Apixaban treatment
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Warfarin Sodium | Apixaban
Number analyzed (Participants) | 13 | 14
percentage of change | -61.45 (43.95) | -65.08 (31.34)

2. Secondary Outcome: Change of Left Ventricular Thrombosis (LVT) by More Than 50%
Description: Percentage of participants who achieved left ventricular thrombus (LVT) reduction more than 50% in both Warfarin and Apixaban arms.
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Warfarin Sodium | Apixaban
Number analyzed (Participants) | 13 | 14
percentage of participants | 77.7 | 61.5

3. Secondary Outcome: Clinically Definite Cardiac Embolic Ischemic Stroke
Description: Number of participants who showed evidence of clinically definite cardiac embolic ischemic stroke (focal neurological deficits persisting for more than 24 hours) confirmed by CT scan
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin Sodium | Apixaban
Number analyzed (Participants) | 13 | 14
Participants | 0 | 1

4. Secondary Outcome: Life Threatening Bleeding
Description: Number of participants who experienced life threatening bleeding attributed to the use of anti-coagulation.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin Sodium | Apixaban
Number analyzed (Participants) | 13 | 14
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Warfarin Sodium | Apixaban
All-Cause Mortality (participants affected / at risk) | 4/13 | 2/14
Serious Adverse Events (participants affected / at risk) | 4/13 | 2/14
Other Adverse Events (participants affected / at risk) | 1/13 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Warfarin Sodium (N=13) | Apixaban (N=14)
Death (Cardiac disorders) | 2 (2) | 1 (1) — Worsening heart failure. Died in hospital.
Gastrointestinal bleeding and Death (Gastrointestinal disorders) | 1 (1) | 0 (0) — Admitted for upper GI bleeding with coagulopathy. Later develop worsening heart failure and died in hospital.
Sudden Death at home (Cardiac disorders) | 1 (1) | 0 (0) — Family informed patient died suddenly at home.
Ischemic Stroke with hemorrhagic transformation and death (Nervous system disorders) | 0 (0) | 1 (1) — Patient develop stroke after off Apixaban 48 hours following end of study. Complicated with hemorrhagic transformation and death.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Warfarin Sodium (N=13) | Apixaban (N=14)
Epistaxis (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Sample size of the study was small due to the pilot nature of the study, being a single-center strict study and strict exclusion criteria.

High rate of early angioplasty in this center also contributed to the low number of patients with left ventricle thrombus (LVT).

Many patients with LVT were excluded because of their ill clinical condition on presentation, deranged renal/liver functions on diagnosis, organized or old LVT and other logistic issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-12-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT02982590/Prot_SAP_ICF_000.pdf